CLINICAL TRIAL: NCT04037891
Title: Topical rVA576 for Treatment of Atopic Keratoconjunctivitis: a Randomised Placebo-controlled Double Masked Parallel Trial (TRACKER)
Brief Title: Topical rVA576 for Treatment of Atopic Keratoconjunctivitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial has terminated early due to the disruptions caused by the ongoing COVID-19 pandemic. The decision was not related to any efficacy, safety or clinical concerns regarding rVA576.
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK701
Record Dates: First submitted 2019-02-13; First posted 2019-07-30 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-07

CONDITIONS: Keratoconjunctivitis, Atopic; Keratoconjunctivitis, Vernal; Conjunctivitis, Allergic
MeSH Terms: conditions — Keratoconjunctivitis; Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomised, double-masked, placebo-controlled parallel group comparison with open-label sentinel group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rVA576 - Open-label period (Experimental): Part 1: The first 3 patients selected for the study will be treated with the active drug in an open-label manner at intervals of 1 week and will have weekly clinic visits until Day 14, after which the visit will be every two weeks. When the first 3 patients have completed two weeks of treatment and the safety and tolerability data has been reviewed by the PI and an independent clinician, provided the data is favourable the randomisation process will begin (Part 2). The first 3 patients will continue treatment for a total of 8 weeks and will be assessed throughout the trial by the Principal Investigator according to the Schedule of Events
  Interventions: Drug: rVA576
- Placebo - Double-blind period (Placebo Comparator): Part 2: Sixteen patients will be randomised 1:1. between active and placebo and patients allocated to either group will receive the appropriate product throughout the trial.
  Interventions: Other: Placebo
- rVA576 - Double-blind period (Experimental): Part 2: Sixteen patients will be randomised 1:1. between active and placebo and patients allocated to either group will receive the appropriate product throughout the trial.
  Interventions: Drug: rVA576

INTERVENTIONS:
Drug: rVA576 — Part 1: The first 3 patients selected for the study will be treated with the active drug in open-label.
  Other Names: Nomacopan
  Arms: rVA576 - Open-label period
Other: Placebo — Part 2: Sixteen patients will be randomised 1:1. between active and placebo and patients allocated to either group will receive the appropriate product throughout the trial.
  Arms: Placebo - Double-blind period
Drug: rVA576 — Part 2: Sixteen patients will be randomised 1:1. between active and placebo and patients allocated to either group will receive the appropriate product throughout the trial.
  Other Names: Nomacopan
  Arms: rVA576 - Double-blind period

SUMMARY:
Topical rVA576 for treatment of atopic keratoconjunctivitis (AKC), vernal keratoconjunctivitis (VKC),and severe allergic conjunctivitis (seasonal (SAC) or perennial (PAC)): a randomised placebo-controlled double masked parallel trial (TRACKER)

DETAILED DESCRIPTION:
Recombinant rVA576 is a small protein (16.7kDa) which has two independent actions. It inhibits the activation and cleavage of complement C5 and it binds and inactivates leukotriene B4 (LTB4). It acts on the complement system by preventing the cleavage of C5 by C5 convertase into C5a and C5b and so is effective in inhibiting terminal complement activity irrespective of the activating pathway.

Atopic keratoconjunctivitis (AKC) is a type of allergic conjunctivitis which involves mast cell activation due to the predominance of inflammatory mediators such as eosinophils and Th2-generated cytokines (Mishra et al. 2011).

Recombinant rVA576 eye drops solution is the investigational medicinal product. It is intended for ophthalmic use by topical administration to the eye.

Recombinant rVA576 is a compact small protein molecule with a lipocalin-like structure consisting of alpha helices and a beta barrel. There is a surface-active site which binds to the complement C5 molecule with a high affinity (KD 1.85 x 10-8 M) and an internalised active site which binds the small eicosinoid molecule leukotriene B4 (Hepburn et al. 2007).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above
2. Diagnosis of moderate to severe AKC, VKC, or severe allergic conjunctivitis (seasonal or perennial). Defined as:

   * AKC, VKC - a composite symptom/sign score from one eye of ≥ 18 out of 33
   * Severe allergic conjunctivitis (SAC or PAC) - a composite symptom/sign score from one eye of ≥ 15 out of 27
3. Will have had received some topical therapy during the last 3 months without improvement but will not currently be receiving systemic immunotherapy. Topical therapy may be topical calcineurin inhibitors, antihistamines or corticosteroids alone or in combination. Lubricants or artificial tears will not a count as topical therapy for these purposes.
4. Will have had at least 7 days without topical ocular corticosteroids prior to entry
5. Willing to give informed consent
6. Willing to use highly effective contraceptive precautions for the duration of the study and for 90 days after the last dose of IMP
7. Willing to avoid prohibited medications for duration of study (see list of prohibited medications)

Exclusion Criteria:

1. Eye surface disease other than AKC, VKC or severe allergic conjunctivitis (SAC or PAC)
2. Contact lens use during the study
3. Complete or partial tarsorrhaphy. If such a procedure becomes necessary during the course of the trial patients may remain in the trial providing that at least 50% of the eye surface remains visible to slit lamp examination
4. Ankyloblepharon of any degree at entry to the trial
5. Known or suspected ocular malignancy
6. Active ocular infection at entry to the trial. Patients with eye surface bacterial, viral, fungal or protozoal infection may enter the trial after elimination of the infection as confirmed by eye swabs
7. Known or suspected uveitis
8. Participation in any other clinical trial within 1 month of enrolment
9. Use of any of the following prohibited medications:

   * Eculizumab
   * Any other investigational complement inhibitor whether systemic or topical (e.g. RA101495)
   * Montelukast
   * Zafirlukast
   * Pranlukast
   * Zileuton
   * Hypericum perforatum (St John's wort)
10. Corneal perforation
11. Uncontrolled glaucoma (increase in dose of glaucoma medication or surgical intervention for glaucoma within 3 months prior to entry)
12. Pregnancy (females)
13. Breast feeding (females)
14. Known allergy to ticks or severe reaction to arthropod venom (e.g. bee or wasp venom)
15. Use of topical ocular steroids within 7 days of the Screening visit
16. Failure to satisfy the PI of suitability to participate for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Ahmad, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (9):
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto Universitario de Oftalmobiología Aplicada, Valladolid
- United Kingdom (7):
  - Bristol Eye Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital NHS Foundation Trust, Southend-on-Sea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in Part 1 did not continue into Part 2.
Groups:
- rVA576, Open-label Period (8 Weeks): Part 1: The first three patients selected were treated with active drug in an open-label manner. They had weekly clinic visits for up the first two weeks and thereafter biweekly visits. When the third of the first three patients had completed their first two weeks of treatment, the PI reviewed the safety, tolerability, and ease of application for each patient before deciding to proceed to the randomised, double masked comparative phase of the study (Part 2). The three patients were to continue on the study and complete eight weeks of treatment as open-label patients.
  Patients in Part 1 did not continue into Part 2.
- rVA576, Double-blind Period (8 Weeks); Placebo (8 Weeks): Part 2: A randomised, double-masked, placebo controlled trial of topical rVA576, or placebo eye drops in moderate to severe AKC, VKC and severe allergic conjunctivitis (SAC or PAC).
Period: Open-label Period
Arm/Group | rVA576, Open-label Period (8 Weeks) | rVA576, Double-blind Period (8 Weeks) | Placebo (8 Weeks)
Started | 3 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Randomized, Double-blind Period
Arm/Group | rVA576, Open-label Period (8 Weeks) | rVA576, Double-blind Period (8 Weeks) | Placebo (8 Weeks)
Started | 0 | 3 (One randomised patient discontinued before receiving the study treatment due to delay in study drug delivery (therefore not included in the number of patients that "Started").) | 6
Completed | 0 | 2 | 6
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- rVA576, Open-label Period: Part 1: The first three patients selected were treated with active drug in an open-label manner. They had weekly clinic visits for up the first two weeks and thereafter biweekly visits. When the third of the first three patients had completed their first two weeks of treatment, the PI reviewed the safety, tolerability, and ease of application for each patient before deciding to proceed to the randomised, double masked comparative phase of the study (Part 2). The three patients were to continue on the study and complete eight weeks of treatment as open-label patients.
- rVA576, Double-blind Period; Placebo: Part 2: A randomised, double-masked, placebo controlled trial of topical rVA576, or placebo eye drops in moderate to severe AKC, VKC and severe allergic conjunctivitis (SAC or PAC).
- Total: Total of all reporting groups
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.55) | 30.3 (6.81) | 33.8 (8.04) | 32.7 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 3 | 2 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Asian | 1 | 1 | 1 | 3
  White | 1 | 1 | 5 | 7
  Other | 1 | 1 | 0 | 2
Indication [Count of Participants; unit: Participants]
  Atopic keratoconjunctivitis (AKC) | 3 | 3 | 2 | 8
  Vernal keratoconjunctivitis (VKC) | 0 | 0 | 2 | 2
  Seasonal allergic conjunctivitis (SAC) | 0 | 0 | 2 | 2
  Perennial allergic conjunctivitis (PAC) | 0 | 0 | 0 | 0
Patient group [Count of Participants; unit: Participants]
  AKC/VKC | 3 | 3 | 4 | 10
  SAC/PAC | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Ocular TEAE
Description: Incidence of ocular treatment-emergent adverse events (TEAE) during the treatment period which have occurred during the 56 days following randomisation.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
Number analyzed (Participants) | 3 | 3 | 6
Participants | 3 | 2 | 3
Statistical Analysis 1: Comparison: rVA576, Double-blind Period vs Placebo; Test type: Superiority; Difference of percentage of participants = 16.7, 95% CI 2-sided [-53.57 to 72.99]
Statistical Analysis 2: Comparison: rVA576, Open-label Period vs rVA576, Double-blind Period vs Placebo; Comparison of incidence of ocular TEAE in all patients receiving rVA576 (part 1 and 2) vs placebo; Test type: Superiority; Difference of percentage of participants = 33.3, 95% CI 2-sided [-25.45 to 78.39]

2. Secondary Outcome: Post-instillation Comfort
Description: Graded on patient diary cards at the intervals Day 1-14, 15-28, 29-42 and 43-56.
  Eye comfort scoring:
  0 - Perfectly comfortable
  1. - Slight discomfort. Some burning, itching or stinging for up to half a minute after using the eye drop, solution but the discomfort improves without treatment.
  2. - Moderate discomfort. Burning, itching or stinging lasts for 0.5 minute or longer but improves without treatment.
  3. - Severe discomfort. Burning, itching or stinging last for at least 0.5 minute and requires washing the eyes to relieve it.
  4. - Unbearable burning itching or stinging. So severe that you cannot continue treatment.
  The 14 day average score for each interval have been calculated for each patient (possible range of 0 to 40). Classifications were assigned using the average total score at each two week period as follows:
  < 10 = Comfortable/Acceptable, 10 - 19 = Moderately Uncomfortable, 20 - 29 = Very Uncomfortable, >= 30 = Severely/Unacceptably Uncomfortable.
Time Frame: Day 1 to 56
Population: The Comfort score data was not available for one patient in the nomacopan group Part 2, and in one patient in Part 1, after Day 14, both due to withdrawal.
  Because only two patients in the Part 2 nomacopan group had data to assess comfort score, it is not meaningful to compare the nomacopan and placebo groups, and so further analysis was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Day 1 to 14: number analyzed (Participants) | 3 | 2 | 6
  Day 1 to 14: Comfortable/Acceptable | 3 | 1 | 4
  Day 1 to 14: Moderately Uncomfortable | 0 | 1 | 2
  Days 15 to 28: number analyzed (Participants) | 2 | 2 | 6
  Days 15 to 28: Comfortable/Acceptable | 2 | 2 | 5
  Days 15 to 28: Moderately Uncomfortable | 0 | 0 | 1
  Days 29 to 42: number analyzed (Participants) | 2 | 2 | 6
  Days 29 to 42: Comfortable/Acceptable | 2 | 1 | 4
  Days 29 to 42: Moderately Uncomfortable | 0 | 1 | 2
  Days 43 to 56: number analyzed (Participants) | 2 | 2 | 6
  Days 43 to 56: Comfortable/Acceptable | 2 | 1 | 5
  Days 43 to 56: Moderately Uncomfortable | 0 | 1 | 1

3. Secondary Outcome: Visual Acuity
Description: Visual acuity for the worst eye over time by Early Treatment Diabetic Retinopathy Study (ETDRS) charts comparison from Day 1 to Day 56 In ETDRS charts, zero indicates standard vision, positive values indicates poor vision, and negative values indicates good vision.
Time Frame: Day 1 to 56
Population: Only one patient in the nomacopan group in Part 2 had data to assess this score. It is not meaningful to compare the nomacopan and placebo groups, and so further analysis was not performed.
Measure: Mean (Standard Deviation); unit: Number of ETDRS letters
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
Number analyzed (Participants) | 3 | 3 | 6
Number of ETDRS letters
  Baseline: number analyzed (Participants) | 3 | 2 | 6
  Baseline | 56.7 (49.1) | 66.0 (19.8) | 82.7 (8.778)
  Day 14: number analyzed (Participants) | 3 | 1 | 6
  Day 14 | 59.0 (48.5) | 82.0 (0) | 82.0 (7.18)
  Day 28: number analyzed (Participants) | 2 | 1 | 6
  Day 28 | 84.0 (0.0) | 78.0 (0) | 79.8 (10.68)
  Day 42: number analyzed (Participants) | 2 | 1 | 4
  Day 42 | 85.5 (0.7) | 83.0 (0) | 79.3 (15.33)
  Day 56 (end of dosing): number analyzed (Participants) | 2 | 1 | 5
  Day 56 (end of dosing) | 87.0 (1.4) | 81.0 (0) | 77.0 (10.56)

4. Secondary Outcome: Clinical Scores
Description: Change from Day 1 in composite clinical scores at Day 14, 28, 42 and 56, for the eye judged as worst affected at each visit. Score calculated from symptom and sign sub-components.
  AKC/VKC: symptom sub-component consisted of itch, tearing, discomfort, discharge, and photophobia, and the sign component consisted of bulbar conjunctival hyperaemia, tarsal conjunctival papillary hypertrophy, punctate keratitis, neovascularization of cornea, cicatrizing conjunctivitis, blepharitis.
  SAC/PAC: symptom sub-component consisted itch, tearing, discomfort, and photophobia, and the sign sub-component consisted of upper tarsal conjunctival hyperaemia, upper bulbar conjunctival hyperaemia, chemosis, upper tarsal conjunctival papillae, blepharitis.
  For each sign/symptom a score of 0 - 3 is awarded (0=absence of a sign/symptom; an increase in score indicates increase in severity). These scores are summed at the end of the exam to give the composite score. Range:0 to 33 (AKC/VKC) or 27 (SAC/PAC).
Time Frame: Day 1 to 56
Population: Because only two patients in the Part 2 nomacopan group had data to assess this score, it is not meaningful to compare the nomacopan and placebo groups, and so further analysis was not performed.
  Note there were two patients on Placebo with SAC; therefore, scored on a different scale compared to patients with AKC or VKC. For the purposes of the outcome measure, the SAC and AKC/VKC scores were combined to derive a single value across all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo (AKC/VKC): Part 2: A randomised, double-masked, placebo controlled trial of topical rVA576, or placebo eye drops in moderate to severe AKC or VKC
- Placebo (SAC/PAC): Part 2: A randomised, double-masked, placebo controlled trial of topical rVA576, or placebo eye drops in moderate to severe AKC, VKC and severe allergic conjunctivitis (SAC or PAC).
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo (AKC/VKC) | Placebo (SAC/PAC)
Number analyzed (Participants) | 3 | 3 | 4 | 2
score on a scale
  Baseline | 23.2 (1.53) | 20.7 (2.31) | 21.3 (1.26) | 19.5 (3.54)
  Day 14: number analyzed (Participants) | 3 | 2 | 4 | 2
  Day 14 | 16.0 (5.20) | 15.0 (1.41) | 14.8 (3.5) | 17.5 (6.36)
  Day 28: number analyzed (Participants) | 2 | 2 | 4 | 2
  Day 28 | 14.5 (0.71) | 19.0 (7.07) | 15 (5.48) | 17.5 (7.78)
  Day 42: number analyzed (Participants) | 2 | 2 | 4 | 0
  Day 42 | 16.0 (7.07) | 16.5 (2.12) | 11.8 (5.32) |
  Day 56: number analyzed (Participants) | 2 | 2 | 4 | 0
  Day 56 | 10.5 (0.71) | 15.0 (1.41) | 11.0 (7.28) |

5. Secondary Outcome: MMP-9 Positive
Description: Percentage of patients with Matrix metalloprotease 9 (MMP-9) positive levels at Days 1, 28, and 56.
  MMP-9 is a is a nonspecific inflammatory marker. Detection was made using the Inflammadry® device. This device gives a binary (positive/negative) result.
Time Frame: Day 1 to 56
Population: There were too few patients to make a meaningful interpretation.
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Baseline left eye: Positive | 2 | 2 | 4
  Baseline left eye: Negative | 1 | 1 | 2
  Baseline right eye: Positive | 2 | 3 | 2
  Baseline right eye: Negative | 1 | 0 | 4
  Day 28 left eye: number analyzed (Participants) | 2 | 2 | 6
  Day 28 left eye: Positive | 0 | 2 | 3
  Day 28 left eye: Negative | 2 | 0 | 3
  Day 28 right eye: number analyzed (Participants) | 2 | 2 | 5
  Day 28 right eye: Positive | 2 | 2 | 2
  Day 28 right eye: Negative | 0 | 0 | 3
  Day 56 left eye: number analyzed (Participants) | 2 | 2 | 5
  Day 56 left eye: Positive | 1 | 1 | 0
  Day 56 left eye: Negative | 1 | 1 | 5
  Day 56 right eye: number analyzed (Participants) | 2 | 2 | 4
  Day 56 right eye: Positive | 1 | 2 | 1
  Day 56 right eye: Negative | 1 | 0 | 3

6. Secondary Outcome: Tear Film Break up Time
Description: Change from Day 1 in Tear film break up time (TBUT) at Day 14, 28, 42 and 56. TBUT data was available for one eye only. Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film. A TBUT under 10 seconds is considered abnormal.
Time Frame: Change from Day 1 at Day 14, 28, 42 and 56
Population: Patient numbers within each treatment group are too small to make meaningful comparisons, and so no further analysis was performed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
Number analyzed (Participants) | 3 | 3 | 6
seconds
  Baseline | 5.0 (5.57) | 3.0 (1.00) | 3.5 (1.05)
  Day 14: number analyzed (Participants) | 3 | 2 | 6
  Day 14 | 6.0 (3.61) | 2.5 (0.71) | 3.7 (2.25)
  Day 28: number analyzed (Participants) | 2 | 2 | 6
  Day 28 | 11.0 (1.41) | 4.5 (0.71) | 5.0 (2.00)
  Day 42: number analyzed (Participants) | 2 | 2 | 4
  Day 42 | 8.0 (0.00) | 4.0 (0.00) | 8.0 (2.16)
  Day 56: number analyzed (Participants) | 2 | 2 | 5
  Day 56 | 6.5 (2.12) | 5.0 (0.00) | 7.4 (1.95)

ADVERSE EVENTS:
Time Frame: From day 1 to day 56.
Arm/Group | rVA576, Open-label Period | rVA576, Double-blind Period | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rVA576, Open-label Period (N=3) | rVA576, Double-blind Period (N=3) | Placebo (N=6)
Atopic keratoconjunctivitis (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Early termination due to the Covid-19 pandemic.
2. Uneven distribution of patients between rVA576 and placebo in Part 2, due to incorrect storage and impossibility of manufacturing a new batch, leading to replacement by the only available randomized and labelled product and resulting in patients being allocated to placebo. With a 6 to 3 distribution of completed patients it is difficult to draw meaningful statistical conclusions or detect trends. The safety data were not compromised.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04037891/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04037891/SAP_001.pdf